CLINICAL TRIAL: NCT02588027
Title: Effect of Ibuprofen on Postoperative Opiate Medication Use and Shoulder Functional Outcomes After Arthroscopic Rotator Cuff Repair
Brief Title: Effect of Ibuprofen on Postoperative Opiate Medication Use and Shoulder Functional Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-16665
Record Dates: First submitted 2015-10-07; First posted 2015-10-27 (Estimated); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Rotator Cuff Tear Arthropathy
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Ibuprofen 400mg by mouth three times daily. Patients will also receive the standard opiate medication (hydrocodone/acetaminophen 10mg/325mg) for the UCSF orthopaedic clinic for postoperative pain control.
  Interventions: Drug: Ibuprofen
- Placebo (Placebo Comparator): Placebo tablet by mouth three times daily. Patients will also received the standard opiate medication (hydrocodone/acetaminophen 10mg/325mg) for the UCSF orthopaedic clinic for postoperative pain control.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibuprofen — Patients will be randomized using a computer generated number to received either ibuprofen (400mg by mouth every eight hours as needed) versus placebo for post-operative pain control in addition to opiate medication (hydrocodone/acetaminophen). Study doctors or research staff will be given randomly generated treatment allocations within sealed opaque envelopes. Once the patient is screened/qualified in surgery, the envelope will be opened and the patient randomized to the allocated treatment regimen. Patients will be given a two week supply (42 pills total) of either ibuprofen or placebo on the day of surgery upon discharge from the surgery center by a research coordinator.
  Other Names: Advil; Motrin
  Arms: Control
Drug: Placebo — Pharmacy formulated placebo
  Arms: Placebo

SUMMARY:
This will be a randomized controlled trial to determine if postoperative ibuprofen after arthroscopic rotator cuff repair impacts postoperative opiate medication use, Visual Analog Scale (VAS) pain scores, shoulder range of motion (ROM), and repair integrity.

DETAILED DESCRIPTION:
Patients will be randomized into two cohorts:

1. Ibuprofen 400mg by mouth three times daily. Patients will also receive the standard opiate medication (hydrocodone/acetaminophen 10mg/325mg) for the UCSF orthopaedic clinic for postoperative pain control.
2. Placebo tablet by mouth three times daily. Patients will also received the standard opiate medication (hydrocodone/acetaminophen 10mg/325mg) for the UCSF orthopaedic clinic for postoperative pain control.

Patients will be screened for the study at the preoperative clinic vist and randomized on the day of surgery if they meet our inclusion criteria.

Postoperatively, they will be seen at 1 week, 6 weeks, 3 months, 6 months, 1 year, and 2 years. Pill counting will be done at the 1 week postoperative visit. VAS pain scores will be assessed at every visit. Functional shoulder outcomes including shoulder range of motion and the American Shoulder and Elbow Society (ASES) survey will be completed at these visits as well. The SF-12 health and Disabilities of Arm, Shoulder, and Hand (DASH) survey will be completed at the preoperative visit and final follow-up visit only. We will assess rotator cuff repair integrity with ultrasound study at 1 year after surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* Patients that undergo arthroscopic rotator cuff repair only

Exclusion Criteria:

* Patients less than 18 years of age, pregnant, are incarcerated. Women who are not post-menopause are screened for pregnancy preoperatively with a urine test per our UCSF Orthopaedic Institute preoperative guidelines.
* Patients who are unable to and not willing to comply with the study protocol and follow-up visits
* Patients with a history of prior rotator cuff repair
* Patients with rotator cuff tears that require open repair
* Patients with an allergy to ibuprofen or anti-inflammatory medications
* Patients with a medical chart record or those who report a history of upper gastroenterology bleed or gastric ulcers
* Patients who are currently on warfarin, enoxaparin, heparin, or a factor Xa inhibiting anti-coagulation medication
* Patients with a known past medical history of chronic kidney disease, history of kidney transplant, or eGFR < 60 mL/min per 1.73m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-10; Primary Completion 2022-09 (Actual); Study Completion 2022-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C. Benjamin Ma, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Orthopaedic Institute, San Francisco, California, United States

REFERENCES:
- [Background] Gilson AM, Ryan KM, Joranson DE, Dahl JL. A reassessment of trends in the medical use and abuse of opioid analgesics and implications for diversion control: 1997-2002. J Pain Symptom Manage. 2004 Aug;28(2):176-88. doi: 10.1016/j.jpainsymman.2004.01.003. PMID 15276196
- [Background] Kang H, Ha YC, Kim JY, Woo YC, Lee JS, Jang EC. Effectiveness of multimodal pain management after bipolar hemiarthroplasty for hip fracture: a randomized, controlled study. J Bone Joint Surg Am. 2013 Feb 20;95(4):291-6. doi: 10.2106/JBJS.K.01708. PMID 23302898
- [Background] Dahl JB, Kehlet H. Non-steroidal anti-inflammatory drugs: rationale for use in severe postoperative pain. Br J Anaesth. 1991 Jun;66(6):703-12. doi: 10.1093/bja/66.6.703. No abstract available. PMID 2064886
- [Background] Dahners LE, Mullis BH. Effects of nonsteroidal anti-inflammatory drugs on bone formation and soft-tissue healing. J Am Acad Orthop Surg. 2004 May-Jun;12(3):139-43. doi: 10.5435/00124635-200405000-00001. PMID 15161166
- [Background] Cohen DB, Kawamura S, Ehteshami JR, Rodeo SA. Indomethacin and celecoxib impair rotator cuff tendon-to-bone healing. Am J Sports Med. 2006 Mar;34(3):362-9. doi: 10.1177/0363546505280428. Epub 2005 Oct 6. PMID 16210573
- [Background] Rouhani A, Tabrizi A, Elmi A, Abedini N, Mirza Tolouei F. Effects of preoperative non-steroidal anti-inflammatory drugs on pain mitigation and patients' shoulder performance following rotator cuff repair. Adv Pharm Bull. 2014 Dec;4(4):363-7. doi: 10.5681/apb.2014.053. Epub 2014 Aug 10. PMID 25436192
- [Background] Tashjian RZ, Deloach J, Porucznik CA, Powell AP. Minimal clinically important differences (MCID) and patient acceptable symptomatic state (PASS) for visual analog scales (VAS) measuring pain in patients treated for rotator cuff disease. J Shoulder Elbow Surg. 2009 Nov-Dec;18(6):927-32. doi: 10.1016/j.jse.2009.03.021. Epub 2009 Jun 16. PMID 19535272
- [Background] van der Zwaal P, Thomassen BJ, Nieuwenhuijse MJ, Lindenburg R, Swen JW, van Arkel ER. Clinical outcome in all-arthroscopic versus mini-open rotator cuff repair in small to medium-sized tears: a randomized controlled trial in 100 patients with 1-year follow-up. Arthroscopy. 2013 Feb;29(2):266-73. doi: 10.1016/j.arthro.2012.08.022. Epub 2012 Dec 1. PMID 23206691

RESULTS

PARTICIPANT FLOW:
Groups:
- Ibuprofen: Ibuprofen 400mg by mouth three times daily. Patients will also receive the standard opiate medication (hydrocodone/acetaminophen 10mg/325mg) for the UCSF orthopaedic clinic for postoperative pain control.
  Ibuprofen: Patients will be randomized using a computer generated number to received either ibuprofen (400mg by mouth every eight hours as needed) versus placebo for post-operative pain control in addition to opiate medication (hydrocodone/acetaminophen). Study doctors or research staff will be given randomly generated treatment allocations within sealed opaque envelopes. Once the patient is screened/qualified in surgery, the envelope will be opened and the patient randomized to the allocated treatment regimen. Patients will be given a two week supply (42 pills total) of either ibuprofen or placebo on the day of surgery upon discharge from the surgery center by a research coordinator.
Period: Overall Study
Arm/Group | Ibuprofen | Placebo
Started | 56 | 54
Completed | 51 | 50
Not Completed | 5 | 4
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Protocol Violation | 4 | 1

BASELINE CHARACTERISTICS:
Population: 110 patients were originally enrolled in the studied however 9 were dropped or elected to withdrawal and did not complete the study medication. Their baseline characteristics were excluded from the analysis because of violation of the protocol or because the patient requested to not have their information as part of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibuprofen | Placebo | Total
Number analyzed (Participants) | 51 | 50 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (10.8) | 56.9 (13.8) | 57.3 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 43
  Male | 29 | 29 | 58
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 32 | 34 | 66
  Hispanic/Latino | 3 | 2 | 5
  Black | 2 | 2 | 4
  Asian | 8 | 8 | 16
  Other | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 51 | 50 | 101
Preoperative NSAID Use [Count of Participants; unit: Participants]
  Ibuprofen | 9 | 8 | 17
  Naproxen | 3 | 3 | 6
  Celecoxib | 0 | 0 | 0
  Other | 1 | 1 | 2
Preoperative Opioid Use [Count of Participants; unit: Participants]
  Norco | 3 | 2 | 5
  Percocet | 0 | 0 | 0
  Oxycodone | 1 | 0 | 1
  Morphine | 0 | 0 | 0
  Hydromorphone | 0 | 0 | 0
Prior Shoulder Cortisone Injection [Count of Participants; unit: Participants] | 15 | 15 | 30
Shoulder Involved [Count of Participants; unit: Participants]
  Right | 27 | 31 | 58
  Left | 24 | 19 | 43
Hand Dominance [Count of Participants; unit: Participants] — Population: Data missing as some patient's did not answer questions regarding hand dominance
  Participants
    Right | 46 | 45 | 91
    Left | 2 | 4 | 6
    Data missing | 3 | 1 | 4
Surgical Side [Count of Participants; unit: Participants] — Population: Some patients did not answer the question regarding hand dominance therefore there are missing data points
  Participants
    Dominant | 24 | 30 | 54
    Non-Dominant | 24 | 19 | 43
    Data missing | 3 | 1 | 4
Size of Rotator Cuff Tear [Count of Participants; unit: Participants] — Population: One patient in the ibuprofen group did not have their tear size categorized by the treating surgeon therefore data point is missing
  Participants
    Small | 21 | 19 | 40
    Medium | 23 | 24 | 47
    Large | 3 | 6 | 9
    Massive | 3 | 1 | 4
    Data missing | 1 | 0 | 1
Tendons Torn [Count of Participants; unit: Participants]
  Supraspinatus | 40 | 42 | 82
  Infraspinatus | 12 | 5 | 17
  Teres Minor | 0 | 0 | 0
  Subscapularis | 25 | 27 | 52
Biceps Tenotomy [Count of Participants; unit: Participants] — Biceps Tenotomy is an additional procedure often performed at the time of rotator cuff surgery if patients have biceps pathology or pain. Documentation of whether not the procedure was performed was based on the surgeon's report and operative note.
  Participants | 6 | 13 | 19
Repair Technique [Count of Participants; unit: Participants] — Single Row and Double Row are surgical repair techniques. Population: repair techniques were not document by the treating surgeon for 5 patients in the ibuprofen group and 3 patients in the placebo group therefore these data points are missing
  Participants
    Single Row | 33 | 33 | 66
    Double Row | 13 | 14 | 27
    Data missing | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Opiate Consumption in Patients Prescribed Ibuprofen Versus Placebo
Description: pain control
Time Frame: 1 week post operative
Measure: Mean (Standard Deviation); unit: morphine milligram equivalents
Arm/Group | Ibuprofen | Placebo
Number analyzed (Participants) | 51 | 50
morphine milligram equivalents | 168.3 (96) | 210.9 (104)

2. Secondary Outcome: Assessment of Functional Shoulder Outcome Score: American Shoulder Elbow Surgery Score (ASES)
Description: American Shoulder Elbow Surgery Score (ASES) - This is a patient reported outcomes score based on a series of questions. The ASES is a 100-point scale that consists of two subscores -- activity of daily living (ADL) and pain visual analog scale (VAS) -- but is reported as one overall score. There is one pain scale worth 50 points and ten activities of daily living worth 50 points. The minimum score is 0 and the maximum score is 100. The higher the score, the better the outcome, indicating better shoulder function (i.e., less pain and better ability to perform daily activities).
Time Frame: Preop, 6-weeks post/op, 3 months post/op, 6 months post/op, 1 year post/op
Population: The number of patients analyzed at the different times points vary from row to row and do not match the overall number of patients in the study due to lost to follow-up of patients over course of study. Several attempts through various means (ie: phone call, email, mail, etc) to reach patients to collect the data were unsuccessful
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ibuprofen | Placebo
Number analyzed (Participants) | 51 | 48
score on a scale
  Preoperative | 57.8 (21.1) | 56.2 (20.7)
  6 weeks: number analyzed (Participants) | 49 | 47
  6 weeks | 54.6 (15.5) | 54 (14.7)
  3 months: number analyzed (Participants) | 45 | 43
  3 months | 69.4 (18.2) | 69.3 (15.9)
  6 months: number analyzed (Participants) | 41 | 39
  6 months | 86.1 (12.1) | 78.1 (17.4)
  1 year: number analyzed (Participants) | 39 | 36
  1 year | 93.4 (8.1) | 90.9 (11.2)

3. Secondary Outcome: Assessment of Functional Shoulder Outcome Score: DASH
Description: The disabilities of the arm, shoulder and hand (DASH) questionnaire is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100. A lower score means a better outcome
Time Frame: preop, 1 year postop
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ibuprofen | Placebo
Number analyzed (Participants) | 50 | 49
score on a scale
  preoperative | 62.6 (20.4) | 62.3 (18.1)
  1 year: number analyzed (Participants) | 41 | 36
  1 year | 31.9 (8.8) | 36.4 (13.6)

4. Secondary Outcome: Assessment of Functional Shoulder Outcome Score: SF-12
Description: The SF-12 (12-item short form health survey) is a general HRQoL survey that measures general health status in 8 domains (physical functioning, role limitations due to physical problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health). Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). Each score ranges from 0 to 100, with higher scores indicating better physical and mental health functioning.
Time Frame: Preop, 1 year post/op
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ibuprofen | Placebo
Number analyzed (Participants) | 50 | 50
score on a scale
  SF-12 PCS preoperative | 42.3 (10.3) | 40.3 (9.4)
  SF-12 PCS 1 year: number analyzed (Participants) | 41 | 37
  SF-12 PCS 1 year | 52.5 (5.8) | 49.4 (9.6)
  SF-12 MCS preoperative | 51.2 (9.5) | 50.1 (11.7)
  Sf-12 MCS 1 year: number analyzed (Participants) | 41 | 37
  Sf-12 MCS 1 year | 53 (9.5) | 51.3 (11.8)

5. Secondary Outcome: Post Operative Pain Score (Visual Analog Scale)
Description: Pain scale from 0 (no pain) - 10 (worst)
Time Frame: 6-weeks post/op, 3 months post/op, 6 months post/op, 1 year post/op
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ibuprofen | Placebo
Number analyzed (Participants) | 49 | 50
score on a scale
  6 weeks | 2.1 (2.0) | 2.5 (2.1)
  3 months: number analyzed (Participants) | 49 | 48
  3 months | 1.8 (1.9) | 1.8 (1.9)
  6 months: number analyzed (Participants) | 41 | 37
  6 months | 0.9 (1.1) | 1.3 (1.5)
  1 year: number analyzed (Participants) | 41 | 36
  1 year | 0.4 (0.8) | 0.7 (1.2)

6. Secondary Outcome: Range of Motion - Forward Flexion
Description: Shoulder motion measured in clinic by a consistent study coordinator/assistant who was blinded to the randomization group using a goniometer. Measurements documented in degrees
Time Frame: Preop, 6-weeks post/op, 3 months post/op, 6 months post/op, 1 year post/op
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Ibuprofen | Placebo
Number analyzed (Participants) | 50 | 50
degrees
  Preoperative | 137 (39) | 133 (40)
  6 weeks: number analyzed (Participants) | 45 | 45
  6 weeks | 92 (29) | 96 (35)
  3 months: number analyzed (Participants) | 43 | 39
  3 months | 142 (19) | 138 (30)
  6 months: number analyzed (Participants) | 40 | 34
  6 months | 162 (14) | 153 (22)
  1 year: number analyzed (Participants) | 42 | 36
  1 year | 168 (16) | 164 (17)

7. Secondary Outcome: Range of Motion - Abduction
Description: as for outcome 6
Time Frame: preoperative, 6 weeks, 3 months, 6 months, 1 year
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Ibuprofen | Placebo
Number analyzed (Participants) | 48 | 50
degrees
  Preoperative | 133 (41) | 125.2 (46)
  6 weeks: number analyzed (Participants) | 45 | 45
  6 weeks | 73 (25) | 76.7 (37)
  3 months: number analyzed (Participants) | 43 | 39
  3 months | 131 (30) | 132.8 (39)
  6 months: number analyzed (Participants) | 40 | 34
  6 months | 164 (21) | 151.6 (33)
  1 year: number analyzed (Participants) | 42 | 36
  1 year | 164 (24) | 161.8 (20)

8. Secondary Outcome: Range of Motion - External Rotation at Side
Description: as for outcome 6
Time Frame: preoperative, 6 weeks, 3 months, 6 months, 1 year
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Ibuprofen | Placebo
Number analyzed (Participants) | 49 | 50
degrees
  preoperative | 58 (18) | 59.7 (18)
  6 weeks: number analyzed (Participants) | 45 | 45
  6 weeks | 35 (13.4) | 36 (17)
  3 months: number analyzed (Participants) | 43 | 39
  3 months | 51 (16) | 56 (17)
  6 months: number analyzed (Participants) | 40 | 34
  6 months | 62 (14) | 57 (18)
  1 year: number analyzed (Participants) | 41 | 36
  1 year | 67 (16) | 65 (17)

9. Secondary Outcome: Range of Motion - External Rotation at 90 Degrees Abduction
Description: as for outcome 6
Time Frame: preoperative, 6 weeks, 3 months, 6 months, 1 year
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Ibuprofen | Placebo
Number analyzed (Participants) | 46 | 48
degrees
  Preoperative | 68 (24) | 68 (29)
  6 weeks: number analyzed (Participants) | 40 | 40
  6 weeks | 42 (18) | 42 (26)
  3 months: number analyzed (Participants) | 42 | 38
  3 months | 69 (16) | 68 (17)
  6 months: number analyzed (Participants) | 40 | 34
  6 months | 78 (13) | 76 (14)
  1 year: number analyzed (Participants) | 42 | 36
  1 year | 83 (12) | 81 (12)

ADVERSE EVENTS:
Time Frame: Data collected for up to 1 year postop
Arm/Group | Ibuprofen | Placebo
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/54
Other Adverse Events (participants affected / at risk) | 0/56 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-09-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT02588027/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT02588027/ICF_001.pdf